CLINICAL TRIAL: NCT01898208
Title: Rapid Identification and Susceptibility Testing of Pathogens Growing in Blood Culture Bottles - A Quality Improvement Theragnostic Stewardship Project
Brief Title: Rapid Identification and Susceptibility Testing of Pathogens From Blood Cultures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Ritu Banerjee, M.D., Ph.D., MD, Ph.D, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11-006920; UM1AI104681 (NIH); KL2TR000136 (NIH)
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Bacteremia; Fungemia; Bloodstream Infection
Keywords: Bacteremia; Fungemia; Bloodstream infection; susceptibility; MRSA; VRE
MeSH Terms: conditions — Bacteremia; Fungemia; Sepsis; Disease Susceptibility | interventions — Antimicrobial Stewardship

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Standard Mayo practices (bacterial culture and susceptibility testing) will be used. FilmArray testing will not be performed.
  Interventions: Other: Bacterial culture; Other: Susceptibility testing
- FilmArray test (Experimental): Standard Mayo practices will be used AND FilmArray testing will be performed. Results of the FilmArray Blood Culture ID Panel test will be communicated to the service by phone in real-time, 24 hours a day, 7 days a week.
  Interventions: Device: FilmArray testing; Other: Bacterial culture; Other: Susceptibility testing
- FilmArray plus antimicrobial stewardship (Experimental): Standard Mayo practices will be used. FilmArray testing will be performed and reported as above, for intervention group 1. IN ADDITION, an expert will review the subject's FilmArray Blood Culture ID Panel result and medical record and contact the primary service if a modification of antimicrobial therapy may be appropriate.
  Interventions: Device: FilmArray testing; Behavioral: Antimicrobial Stewardship; Other: Bacterial culture; Other: Susceptibility testing

INTERVENTIONS:
Device: FilmArray testing — FilmArray Blood Culture Identification (BCID) Panel is a polymerase chain reaction (PCR) panel that identifies 19 types of bacteria, 5 types of fungi, and select antimicrobial-resistance genes.
  Other Names: FilmArray Blood Culture Identification Panel
  Arms: FilmArray plus antimicrobial stewardship; FilmArray test
Behavioral: Antimicrobial Stewardship — Real time antimicrobial stewardship: an infectious diseases pharmacist or physician will provide patient-specific recommendations to modify antimicrobial therapy.
  Arms: FilmArray plus antimicrobial stewardship
Other: Bacterial culture — This test identifies the pathogen responsible for an infection.
Other: Susceptibility testing — Antibiotic susceptibility testing determines the susceptibility of a bacterial strain to a specific antibiotic or a panel of antibiotics. Antibiotic susceptibility testing determines the susceptibility of a bacterial strain to a specific antibiotic or a panel of antibiotics.

SUMMARY:
Would rapid identification of bacteria and rapid detection of methicillin-resistant S. aureus (MRSA) and vancomycin-resistant enterococci (VRE) (using an FDA-cleared assay) in positive blood culture bottles improve patient care at Mayo Clinic Rochester (or just lead to increased cost)?

DETAILED DESCRIPTION:
We hypothesize that the FilmArray Blood Culture ID Panel will reduce the duration of empiric broad-spectrum antimicrobial therapy typically administered in patients who have positive blood cultures, improving clinical outcome and reducing cost. To test this hypothesis we propose a prospective, randomized controlled study comparing outcomes among patients with positive blood cultures who receive either: Standard culture and antimicrobial susceptibility testing (AST) of positive blood culture bottles as is done today (control), standard culture and AST of positive blood culture bottles plus the FilmArray Blood Culture ID Panel (intervention group 1), or standard culture and AST of positive blood culture bottles plus the FilmArray Blood Culture ID Panel testing along with expert infectious diseases phone consultation (intervention group 2). In both intervention groups, results of the FilmArray test will be communicated by phone to the primary service, along with templated comments about optimal antimicrobial therapy, based on the result. (Templated comments will also be used in the control group). In intervention group 2, an infectious diseases pharmacist or physician will provide patient-specific recommendations to modify antimicrobial therapy, if appropriate, based on microbiology results and clinical information obtained through medical record review and discussion with the primary service.

ELIGIBILITY:
Inclusion criteria:

* Positive blood culture during the study period.
* No positive blood cultures in prior 7 days
* Minnesota state research authorization provided

Exclusion criteria:

* No Minnesota state research authorization
* Deceased or transitioned to comfort care within 24 hours of enrollment
* Positive blood culture in prior 7 days
* Previously enrolled in this study
* Negative Gram stain

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Patel, MD, Principal Investigator — Mayo Clinic; Ritu Banerjee, MD, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banerjee R, Teng CB, Cunningham SA, Ihde SM, Steckelberg JM, Moriarty JP, Shah ND, Mandrekar JN, Patel R. Randomized Trial of Rapid Multiplex Polymerase Chain Reaction-Based Blood Culture Identification and Susceptibility Testing. Clin Infect Dis. 2015 Oct 1;61(7):1071-80. doi: 10.1093/cid/civ447. Epub 2015 Jul 20. PMID 26197846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic in Rochester, Minnesota from August 2013 to March 2014.
Groups:
- Control: Standard Mayo practices (culture and susceptibility testing) will be used. FilmArray testing will not be performed.
- FilmArray Test: Standard Mayo practices will be used AND FilmArray testing will be performed. Results of the FilmArray Blood Culture Infectious Disease (ID) Panel test will be communicated to the service by phone in real-time, 24 hours a day, 7 days a week.
Period: Overall Study
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Started | 247 | 247 | 249
Completed | 207 | 198 | 212
Not Completed | 40 | 49 | 37
Not completed — Positive blood culture | 17 | 23 | 15
Not completed — Death/comfort care within 24 hours | 10 | 9 | 8
Not completed — Negative Gram Stain | 6 | 9 | 6
Not completed — Non-Blood Specimens in Bottles | 3 | 5 | 4
Not completed — System/Technical Error | 1 | 2 | 3
Not completed — Lost to Follow-up | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized subjects were excluded if they had a positive blood culture in the prior week, had not provided the state research authorization, previously enrolled in the study, died or transitioned to comfort care within 24 hours of enrollment, or had a negative Gram stain. Only non-excluded subjects were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship | Total
Number analyzed (Participants) | 207 | 198 | 212 | 617
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (19.32) | 61.4 (21.22) | 61.2 (20.08) | 61.4 (20.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 82 | 85 | 232
  Male | 142 | 116 | 127 | 385
Region of Enrollment [Number; unit: participants]
  United States | 207 | 198 | 212 | 617

OUTCOME MEASURES:

1. Primary Outcome: Duration of Antimicrobial Therapy (Hours)
Description: Difference between the date and time of the antibiotic start order (or Gram stain-positive blood culture, if antibiotics were started prior to the positive culture result) and the date and time of the antibiotic stop order. Shorter duration of broad spectrum antibiotics and longer duration of narrow-spectrum antibiotics were considered favorable outcomes.
Time Frame: Approximately 4 days after enrollment
Population: Subjects could have received more than one antimicrobial. Participants analyzed per variable below are expressed as (n=control, FilmArray test, and FilmArray+Stewardship)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
hours
  Vancomycin (van), all subjects (n=132, 101, 124) | 44 [22 to 72] | 42 [21 to 93] | 42 [19 to 90]
  Van, organisms not requiring van (n=56, 56,57) | 8.2 [0 to 26] | 0 [0 to 16] | 0 [0 to 3]
  Van-susceptible enterococci (n=8, 8, 16) | 20 [1 to 59] | 70 [48 to 88] | 82 [40 to 96]
  Van, Methicillin-susceptible S.aureus(n=13,13,16) | 23 [20 to 53] | 11 [0 to 26] | 8 [0 to 44]
  Nafcillin, oxacillin, or cefazolin (n=20, 16, 14) | 42 [24 to 57] | 71 [51 to 79] | 85 [42 to 92]
  Piperacillin-tazobactam (n=77, 65, 72) | 56 [39 to 82] | 44 [27 to 74] | 45 [19 to 78]
  Cefepime (n=62, 52, 67 | 55 [28 to 96] | 71 [43 to 96] | 58 [32 to 96]
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For Vancomycin, all patients; Test type: Superiority or Other; p = 0.92, Kruskal-Wallis
Statistical Analysis 2: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For vancomycin, organisms not requiring vancomycin; Test type: Superiority or Other; p = 0.032, Kruskal-Wallis
Statistical Analysis 3: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For vancomycin-susceptible enterococci; Test type: Superiority or Other; p = 0.037, Kruskal-Wallis
Statistical Analysis 4: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For vancomycin, methicillin-susceptible Staphylococcus aureus; Test type: Superiority or Other; p = 0.2, Kruskal-Wallis
Statistical Analysis 5: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For nafcillin, oxacillin, or cefazolin; Test type: Superiority or Other; p = 0.035, Kruskal-Wallis
Statistical Analysis 6: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For piperacillin-tazobactam; Test type: Superiority or Other; p = 0.012, Kruskal-Wallis
Statistical Analysis 7: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For cefepime; Test type: Superiority or Other; p = 0.56, Kruskal-Wallis

2. Secondary Outcome: Time From Positive Gram Stain to First Active Antibiotic
Description: From positive Gram stain to start of active antibiotic among patients not on active therapy at enrollment; excludes subjects with contaminated blood cultures.
Time Frame: Approximately 14 days after positive blood culture
Population: Not all subjects were not on active therapy at enrollment, and also subjects with contaminated blood cultures were excluded. Participants analyzed per variable below are expressed as (n=control, FilmArray test, and FilmArray+Stewardship): (n=45, 41, 37)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
hours | 11 [2 to 51] | 6 [2 to 31] | 4 [2 to 20]
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; This analysis compares the 3 groups; Test type: Superiority or Other; p = 0.55, Kruskal-Wallis

3. Secondary Outcome: Time to First Appropriate De-escalation or First Appropriate Escalation of Antibiotics
Description: De-escalation included discontinuation of 1 or more antibiotics and/or switching from a broad- to a narrow spectrum antibiotic. Escalation included initiation of 1 or more antibiotics and/or switching from a narrow- to a broad-spectrum antibiotic.
Time Frame: Positive Gram stain, 96 hours after enrollment
Population: Not all subjects experienced de-escalation or escalation of their antibiotics. Participants analyzed per variable below are expressed as (n=control, FilmArray test, and FilmArray+Stewardship).
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 247 | 249
hours
  Time to first approp. de-escalation(n=121,112,111) | 34 [21 to 55] | 38 [22 to 66] | 21 [7 to 37]
  Time to first appropriate escalation (40,38,44) | 24 [3 to 67] | 6 [2 to 36] | 5 [2 to 22]
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For time to first appropriate de-escalation comparing the 3 groups; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; For time to first appropriate escalation comparing the 3 groups; Test type: Superiority or Other; p = 0.04, Kruskal-Wallis

4. Secondary Outcome: Percent of Contaminated Blood Cultures Not Treated or Treated for Less Than 24 Hours
Description: Contaminated blood cultures were defined as growth of organisms such as coagulase-negative staphylococci from a single blood culture set when greater than or equal to 2 blood culture sets were collected, except among subjects suspected to have true bacteremia associated with central venous catheters or devices.
Time Frame: Within 14 days after positive blood culture
Measure: Number; unit: Percentage of blood cultures
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
Percentage of blood cultures | 75 | 89 | 92
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; This analysis compares the 3 groups; Test type: Superiority or Other; p = 0.015, Chi-squared

5. Secondary Outcome: Time to Pathogen Identification
Time Frame: Approximately 14 days after positive blood culture
Population: The number of subjects analyzed per arm differs from the number of subjects who completed the study because this outcome measure includes only the subset of subjects who had organisms represented on the rapid multiplex PCR (rmPCR) panel.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 169 | 147 | 165
hours | 22.3 [17 to 28] | 1.3 [0.9 to 1.6] | 1.3 [0.9 to 1.6]
Statistical Analysis 1: Comparison: Control vs FilmArray Test; This analysis compares the FilmArray test to control arm; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Control vs FilmArray Plus Antimicrobial Stewardship; This analysis compares FilmArray plus antimicrobial stewardship to the control arm; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis

6. Secondary Outcome: Number of Subjects Who Had Negative Blood Cultures Within 3 Days After Enrollment
Time Frame: 3 Days after enrollment
Measure: Number; unit: participants
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
participants | 147 | 131 | 146
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; This analysis is to compare the three groups; Test type: Superiority or Other; p = 0.79, Kruskal-Wallis

7. Other Pre Specified Outcome: Length of Intensive Care Unit Stay
Time Frame: within 14 days of positive blood culture until ICU discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
days | 3 [2 to 4] | 2 [1 to 5] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; Test type: Superiority or Other; p = 0.90, Kruskal-Wallis

8. Other Pre Specified Outcome: Percentage of Patients Who Acquired Clostridium Difficile or Multidrug-resistant Organisms Within 30 Days After Enrollment
Description: Multidrug-resistant organisms included vancomycin-resistant enterococci, methicillin-resistant Staphylococcus aureus, extended-spectrum cephalosporin-resistant Enterobacteriaceae, and Pseudomonas aeruginosa and Acinetobacter species resistant to greater than or equal to 3 antibiotic classes.
Time Frame: Approximately 30 days after positive blood culture
Measure: Number; unit: percentage of participants
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
percentage of participants | 7.2 | 8.1 | 9.9
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; This analysis is a comparison of the 3 groups; Test type: Superiority or Other; p = 0.62, Chi-squared

9. Secondary Outcome: Length of Entire Hospitalization (Days)
Time Frame: Participants were followed for the duration of hospital stay, approximately 15 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
days | 8 [5 to 15] | 8 [5 to 15] | 8 [5 to 16]
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; This analysis compares the three groups; Test type: Superiority or Other; p = 0.60, Kruskal-Wallis

10. Secondary Outcome: All-cause and Attributable Mortality
Description: If records of death were incomplete, mortality was determined using Accurint (LexisNexis, Philadelphia, PA), an internet research and location service.
Time Frame: 30 days after positive blood culture
Measure: Number; unit: participants
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
participants
  All-cause mortality | 22 | 20 | 18
  Attributable mortality | 7 | 7 | 2
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; Comparison of the 3 groups for all-cause mortality; Test type: Superiority or Other; p = 0.74, Fisher Exact
Statistical Analysis 2: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; Comparison of the 3 groups for attributable mortality; Test type: Superiority or Other; p = 0.42, Fisher Exact

11. Secondary Outcome: Number of Subjects With Antibiotic-Associated Toxicities/Adverse Events
Description: This included all adverse events that occurred within 2 weeks following enrollment and were documented in the medical record.
Time Frame: Approximately 14 days after positive blood culture
Measure: Number; unit: participants
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
participants | 3 | 3 | 2
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; This analysis is a comparison across all three groups; Test type: Superiority or Other; p = 0.82, Fisher Exact

12. Secondary Outcome: Percentage of Subjects With Infectious Disease Consultation Within 72 Hours of Enrollment
Time Frame: Approximately within 72 hours of positive blood culture
Measure: Number; unit: percentage of participants
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 207 | 198 | 212
percentage of participants | 49.8 | 49 | 45.3

13. Secondary Outcome: Mean Total Hospitalization, Laboratory Test, and Antimicrobials Costs Per Subject
Description: Costs were calculated using a standardized inflation-adjusted estimate of costs for each service or procedure performed in constant dollars. This approach adjusts for hospital-billed charges with Medicare Cost Report department-level cost-to-charge ratios. Physician services were proxied with Medicare reimbursement rates based on Current Procedure Terminology (CPT)-4 codes using the Medicare Fee Schedule. We did not include the cost of the stewardship program in the cost analysis, as it is not a billed service. As there was no Medicare reimbursement rate for the rmPCR test at the time of the study, test cost was proxied using the FilmArray respiratory panel. These costs were varied in sensitivity analysis with rmPCR test cost ranging from a 50% decrease to a 300% increase.
Time Frame: Approximately 7 days after positive blood culture and for duration of entire hospitalization
Population: The number of subjects analyzed per arm is different than the number of subjects who completed the study because outpatients and a few subjects without final billing data available were excluded.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Number analyzed (Participants) | 191 | 171 | 182
dollars
  Overall Hospitalization Costs | 65,450 (128,686) | 66,887 (117,832) | 68,729 (134,215)
  Laboratory Test Cost | 5,377 (10,115) | 5,680 (8,872) | 5,743 (9,809)
  Antimicrobials Costs | 2,194 (4,175) | 1,932 (3,175) | 1,741 (2,748)
Statistical Analysis 1: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; Comparison between the 3 arms for total hospitalization costs; Test type: Superiority or Other; p = 0.7789, Kruskal-Wallis
Statistical Analysis 2: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; Comparison between the 3 arms for laboratory test cost; Test type: Superiority or Other; p = 0.0006, Kruskal-Wallis
Statistical Analysis 3: Comparison: Control vs FilmArray Test vs FilmArray Plus Antimicrobial Stewardship; Comparison between the 3 arms for antimicrobials costs; Test type: Superiority or Other; p = 0.6540, Kruskal-Wallis

ADVERSE EVENTS:
Description: All events that occurred within 2 weeks following enrollment and were documented in the medical record were collected.
Arm/Group | Control | FilmArray Test | FilmArray Plus Antimicrobial Stewardship
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/198 | 0/212
Other Adverse Events (participants affected / at risk) | 3/207 | 3/198 | 2/212
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=207) | FilmArray Test (N=198) | FilmArray Plus Antimicrobial Stewardship (N=212)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myelosuppression (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes